CLINICAL TRIAL: NCT06906016
Title: New Biomarkers of HBV Infection: Clinico-Biological Characterization and Impact on Infection Management
Brief Title: New HBV Infection Biomarkers: Clinical Characterization and Impact on Management
Acronym: HBV-Biomark
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230425
Record Dates: First submitted 2025-03-04; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Chronic Hepatitis B Virus (HBV) Infection
Keywords: Chronic Hepatitis B (HBV); HBV RNA; HBV biomarkers; Hepatocellular carcinoma (HCC); HBV genotyping; Hepatitis B treatment
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B; Infections; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples: Collected during the regular medical consultations of the patients. These samples will be used to assess various biomarkers associated with the HBV infection.
  Research-specific samples:
  9 mL of dry tube (serum): This sample will be used for analyzing various biomarkers, including the quantification of viral RNA, and assessing other clinical markers of HBV infection.
  9 mL Paxgene tube: This sample will be used for RNA extraction, which is crucial for studying the virus's RNA (HBV RNA) and its role in viral replication, as well as other potential molecular characteristics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort Study on Chronic HBV Infection: This study is a cohort study. It follows a group of patients infected with HBV (Hepatitis B) over an extended period to evaluate the predictive role of biomarkers in the progression of the infection and the response to antiviral treatment. Patients are monitored over time, with regular sample collection to measure biomarkers and assess clinical and biological events, such as seroconversion or the emergence of complications like cirrhosis or liver cancer.
  Interventions: Biological: Collection of blood samples for the study of HBV biomarkers

INTERVENTIONS:
Biological: Collection of blood samples for the study of HBV biomarkers — The intervention involves the additional and minimal collection of two blood samples during routine care procedures (9mL in a dry tube and 9mL in a Paxgene tube). These samples are specifically collected for research purposes and will be stored in the laboratory at the Henri Mondor Biobank Platform under the responsibility of Pr Bijan Ghaleh-Marzban for 15 years. The samples will be preserved under strict conditions and may be used for future analyses related to the pathology of HBV infection or other scientific advancements, with the patient's informed consent.

SUMMARY:
Chronic Hepatitis B Virus (HBV) infection affects nearly 300 million people worldwide and is a leading cause of liver fibrosis, cirrhosis, and hepatocellular carcinoma (HCC). In France, it affects around 0.3% of the population. Current clinical practice relies on traditional biomarkers, such as HBV DNA and HBsAg, to monitor viral replication and disease progression. However, these biomarkers do not fully capture the viral activity or predict clinical outcomes. Recently, new biomarkers like HBcrAg and HBV RNA have emerged, showing promise for better understanding the natural history of the infection and guiding treatment decisions. The main objective of this research is to evaluate the predictive role of these biomarkers (HBcrAg, HBV RNA) in HBV-infected patients, focusing on their association with HBsAg seroconversion and their ability to predict clinical events like cirrhosis and HCC. Secondary objectives include describing the clinicobiological characteristics of patients, determining HBV genotypes, characterizing the impact of HBV on the host's transcriptome, and studying the biomarkers' role in different phases of the infection and treatment. The ultimate goal is to identify more accurate biomarkers to guide antiviral treatment, predict disease progression, and potentially determine when treatment can be safely discontinued.

DETAILED DESCRIPTION:
This study focuses on the chronic Hepatitis B virus (HBV) infection, which affects nearly 300 million people globally, leading to cirrhosis, hepatocellular carcinoma (HCC), and other severe liver diseases. The objective is to evaluate new biomarkers for HBV infection, specifically HBV core-related antigen (HBcrAg) and HBV RNA, and their potential role in the clinical management and prognosis of the disease. Traditional biomarkers used to track viral replication and liver fibrosis, such as HBV DNA, HBeAg, and HBsAg, have limitations, which this study aims to address by exploring emerging biomarkers that could improve the understanding of the infection's natural history and response to antiviral treatments.

The population involved in the study includes patients diagnosed with chronic HBV infection and receiving care at Henri Mondor-Albert Chenevier University Hospital. Patients must be 18 years or older and have been infected with HBV (positive HBsAg for more than six months). Exclusion criteria include individuals with liver transplantation history, those unable to provide consent, pregnant or breastfeeding women, and those not affiliated with a Social Security scheme.

The study design includes both primary and secondary evaluation criteria. The primary criterion is the incidence of HBsAg seroconversion (absence of detectable HBsAg in serum). Secondary criteria include the proportion of patients positive for HBeAg, the incidence of clinical events like cirrhosis and HCC, and the molecular characterization of HBV, such as genotype distribution and the presence of co-infections like hepatitis C (HCV) or HIV. Other secondary criteria also include the measurement of liver fibrosis using Fibroscan and screening for HCC through abdominal ultrasound and alpha-fetoprotein (AFP) tests.

Research procedures involve routine medical consultations, with additional blood samples (9mL dry tube and 9mL Paxgene) collected for research purposes once a year. Patients will be followed for a period of 10 years, with regular monitoring of HBV biomarkers and liver status to evaluate the progression of the infection, the risk of developing liver disease, and the potential predictive value of new biomarkers for viral replication and clinical outcomes. The ultimate aim is to enhance HBV management by identifying predictive biomarkers and refining treatment strategies, particularly to optimize antiviral therapies and improve patient prognosis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* Chronic HBV infection (HbsAg positive carrier for more than 6 months)
* Patient under care within the Henri Mondor-Albert Chenevier University Hospital group

Exclusion Criteria:

* History of liver transplantation for liver failure in the context of chronic HBV infection
* Protected adults, adults unable to express their consent
* Pregnant or breastfeeding women
* Person not affiliated with a Social Security system
* Patient refusal to participate in the project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients infected with HBV, followed in the hepatology department - Henri-Mondor University Hospital.
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2038-11-27 (Estimated); Study Completion 2038-11-27 (Estimated)

PRIMARY OUTCOMES:
HBsAg Seroconversion Rate | 3 months
  Defined by the absence of detectable AgHBs in the serum using ELISA test

SECONDARY OUTCOMES:
Incidence of Biological Events | 1 year
  Monitoring the seroconversion of HBeAg using biological data, measured by the proportion of patients with HBeAg seroconversion.
Quantification of VHB Transcripts | 1 year
  Quantitative analysis of VHB transcripts using PCR, measured in copies per milliliter (copies/ml).
Biomarker Quantification: VHB RNA | 1 year
  Quantification of the virus biomarker VHB RNA during follow-up using PCR, measured in copies per milliliter (copies/ml).
Diagnosis of Liver Tumor | 1 year
  Diagnostic assessment of liver tumors using medical imaging techniques, such as MRI
Incidence of Clinical Events | 1 year
  Monitoring of clinical events, such as cirrhosis, measured by the proportion of patients affected by clinical events.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Unit (CRU) Henri Mondor., Créteil, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION